CLINICAL TRIAL: NCT04575103
Title: Monitoring of Arrhythmias in Patients Treated With Antipsychotics - The MAPP II Study
Brief Title: Monitoring of Arrhythmias in Patients Treated With Antipsychotics
Acronym: MAPP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Herlev and Gentofte Hospital (Other)
Collaborators: Rigshospitalet, Denmark (Other); Bispebjerg Hospital (Other); Nordsjaellands Hospital (Other); University Hospital, Gentofte, Copenhagen (Other); Zealand University Hospital (Other); Odense University Hospital (Other); Aarhus University Hospital (Other); Aalborg University Hospital (Other)
Responsible Party: Principal Investigator, Casper N. Bang, Principal Investigator, University Hospital Bispebjerg and Frederiksberg
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: A0001
Record Dates: First submitted 2020-09-24; First posted 2020-10-05 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Death, Sudden, Cardiac; Arrythmia; Antipsychotics and Neuroleptics Toxicity
MeSH Terms: conditions — Death, Sudden, Cardiac; Arrhythmias, Cardiac | interventions — Antipsychotic Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Antipsychotics (Active Comparator): Patients treated with antipsychotics as provided by their psychiatrist in order to treat disease best possible and in accordance with guidelines.
  Interventions: Drug: Antipsychotic
- Control (No Intervention): Healthy controls, not treated with antipsychotics.

INTERVENTIONS:
Drug: Antipsychotic — Antipsychotic treatment >0.5 DDD
  Arms: Antipsychotics

SUMMARY:
Antipsychotics may be associated to life-threatening arrhythmias and sudden cardiac death. This is the fist study to estimated the arrhythmic burden using long-term monitoring by implantable loop recorder in patients treated with antipsychotics.

DETAILED DESCRIPTION:
Aims and objectives To estimate frequency of potential malign arrhythmias and cardiovascular outcome in a population with patients treated with antipsychotic drugs compared to healthy controls.

Background Life expectancy is about 20 years shorter for patients with mental illness compared to the general population. Increasing evidence suggest that antipsychotic drugs can cause cardiac arrhythmias and hence sudden death. However, the evidence as well as the incidence of rhythm disturbances in patients treated with antipsychotic drugs is insufficient reported. Prolonged monitoring with external portable monitors is difficult for practical and technical reasons. In addition, long-term consistent and structured timing of clinical visits is often a challenge in this vulnerable patient group. In recent years, patients who have been suspected of rarely occurring arrhythmias, have been offered long-term monitoring using an 'implantable loop recorder' (ILR). However, no study has evaluated the arrhythmic burden in patients treated with antipsychotic drugs using ILR.

Methods and materials The study is a national joint project between departments of psychiatry and cardiology across Denmark. After written informed consent and a baseline evaluation including echocardiography, ecg and biochemistry, an ILR will be implanted. During follow-up, arrhythmias will be monitored at regular clinical visits. Cardiovascular endpoints will be monitored using Danish national registries.

Expected outcome and perspectives The present study is the first to reveal arrhythmias among patients treated with antipsychotics using consistent long-term monitoring. The results will give valuable insights into possible mechanism of the observed early death and risk of sudden death in patients treated with antipsychotics.

ELIGIBILITY:
Inclusion Criteria:

* Patients with SMI defined according to ICD-10 as:

  * F20.0-F20.9 schizophrenia
  * F22.0-F22.9 paranoid psychosis
  * F25.0-F25.9 schizo-affective psychosis
  * F28 other non-organic psychosis
  * F29 non-organic psychosis unspecified
  * F31.0-F31.9 bipolar affective disorder.
* Patients treated with or initiating antipsychotics with ≥ 0.5 daily defined dosage
* >18 years old and <50 years.

Exclusion Criteria:

* Patients not capable to understand the aim of the study as judged by investigator.
* Current in treatment with methadone.
* Left ventricular hypertrophy (echocardiographic septal thickness ≥1.3 cm for women and ≥1.4 cm for men, or LVM/BSA ≥109 g/m2 for women or ≥132 g/m2 for men).
* Heart failure (echocardiographic LVEF <35%).
* Ischemic heart disease (patient reported coronary bypass grafting or percutaneous coronary intervention.
* Congenital cardiovascular disease (patient reported).

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 600 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Ventricular arrhythmias | 2 years from insertion og loop recorder
  Number of patients with ventricular arrhythmias detected on insertable loop recorder

SECONDARY OUTCOMES:
Supraventricular arrhythmias | 2 years from insertion og loop recorder
  Number of patients with supraventricular arrhythmias including atrial fibrillation or flutter detected on insertable loop recorder.
Bradycardia | 2 years from insertion og loop recorder
  Number of patients with bradycardia (defined as resting rate lower than 40/min) detected on insertable loop recorder.

OTHER OUTCOMES:
Long QT interval | 2 years from insertion og loop recorder
  Number of patients with long QT interval on routine ECG or detected on insertable loop recorder defined as QTc > 500 ms.
Pacemaker/ICD implantation. | 2 years from insertion og loop recorder
  Number of patients who receives pacemaker/ICD implantation using questionnaire and national pace- and ICD register.
Sudden cardiac death. | 2 years from insertion og loop recorder
  Number of patients who experiences sudden cardiac death using national death and diagnosis register.
Cardiovascular mortality | 2 years from insertion og loop recorder
  Number of patients who experiences cardiovascular mortality using national death and diagnosis register.
All-cause mortality | 2 years from insertion og loop recorder
  Number of patients who experiences all-cause mortality using national death and diagnosis register.
Suicide or death caused by non-cardiac factors | 2 years from insertion og loop recorder
  Number of patients who experiences suicide or death caused by non-cardiac factors using national death and diagnosis register.
Frequency of primary endpoint in controls | 2 years from insertion og loop recorder
  Frequency of primary endpoint in controls detected on insertable loop recorder.
Frequency of primary endpoint related to specific psychiatric drugs / dose | 2 years from insertion og loop recorder
  Frequency of primary endpoint related to specific psychiatric drugs / dose detected on insertable loop recorder
Frequency of primary endpoint related to the presence of long QTc interval | 2 years from insertion og loop recorder
  Frequency of primary endpoint related to the presence of long QTc interval detected on insertable loop recorder
Frequency of primary endpoint in poor metabolizers compared to normal metabolizers | 2 years from insertion og loop recorder
  Frequency of primary endpoint in poor metabolizers compared to normal metabolizers detected on insertable loop recorder
Frequency of primary endpoint by genetic analysis | 2 years from insertion og loop recorder
  Frequency of primary endpoint by genetic analysis detected on insertable loop recorder.

CONTACTS AND LOCATIONS:
Overall Officials: Casper Bang, MD, PhD, Principal Investigator — Department of Cardiology, Bispebjerg and Frederiksberg Hospital, Copenhagen University, Denmark
Locations (18):
- Denmark (18):
  - Department of Psychiatry, Region of Southern Denmark, Aabenraa
  - Cardiology, Aalborg Universitetshospital, Aalborg
  - Psychiatry, Aalborg University Hospital, Aalborg
  - Aarhus Universitetshospital, Skejby, Department of Cardiology, Aarhus
  - Department of Psychiatry, Aarhus University, Aarhus
  - Bispebjerg Hospital, Department of Cardiology, Copenhagen
  - Copenhagen Center of Psychiatry (Rigshospitalet), Copenhagen
  - Mental Health Center Amager, Copenhagen
  - Rigshospitalet, Department of Cardiology, Copenhagen
  - Mental Health Center Frederiksberg, Frederiksberg
  - Gentofte-Herlev Hospital, Department of Cardiology, Gentofte Municipality
  - Mental Health Center Glostrup, Glostrup Municipality
  - Mental Health Center Copenhagen, Hellerup
  - North Zealand Hospital, Department of Cardiology, Hillerød
  - North Zealand Hospital, Department of Psychiatry, Hillerød
  - Odense University Hospital, Department of Cardiology, Odense
  - Zealand University Hospital, Department of Cardiology, Roskilde
  - Psychiatric Research Unit, Region of Zealand, Slagelse

IPD SHARING:
Plan to Share IPD: No